CLINICAL TRIAL: NCT00528996
Title: A Multinational, Randomised, Double-blind, Placebo- and Active-controlled, Parallel Group Efficacy and Safety Comparison Over 24 Weeks of Three Doses (50µg, 100µg, 200µg) of BEA 2180 BR to Tiotropium 5µg, Delivered by the Respimat Inhaler and Placebo in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: An Efficacy and Safety Study to Compare Three Doses of BEA 2180 BR to Tiotropium and Placebo in the Respimat Inhaler.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1205.14; 2007-007946-42
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo
- BEA 2180 BR low dose (Experimental): Low dose
  Interventions: Drug: BEA 2180 BR
- BEA 2180 BR medium dose (Experimental): Medium dose
  Interventions: Drug: BEA 2180 BR
- BEA 2180 BR high dose (Experimental): High dose
  Interventions: Drug: BEA 2180 BR
- Tiotropium Bromide (Experimental): Tiotropium Bromide
  Interventions: Drug: Tiotropium Bromide

INTERVENTIONS:
Drug: BEA 2180 BR — Solution
  Arms: BEA 2180 BR high dose; BEA 2180 BR low dose; BEA 2180 BR medium dose
Drug: Tiotropium Bromide — Solution
  Arms: Tiotropium Bromide
Drug: Placebo — Solution
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the bronchodilator efficacy of three doses (50 µg, 100 µg and 200 µg) of BEA 2180 delivered by the Respimat® once daily to placebo and tiotropium bromide delivered by the Respimat® in patients with COPD. Additional objectives include comparing the effects on dyspnea and health status.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease (P95 4381) and must meet the following spirometric criteria:

   Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 (post-bronchodilator, 30 minutes post salbutamol/albuterol) <80% of predicted normal and FEV1 less than or equal to 70% of FVC at the PFTs at Visit 1 (screening).
3. Male or female patients 40 years of age or older.
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years. Patients who have never smoked cigarettes must be excluded.
5. Patients must be able to perform technically acceptable pulmonary function tests and electronic PEFR measurements, and must be able to maintain records (Patient Daily Diary) during the study period as required in the protocol.
6. Patients must be able to inhale medication in a competent manner from the Respimat® inhaler (Appendix I)

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient ability to participate in the study.
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defines a significant disease as defined in exclusion criterion No. 1.
3. Patients with a recent history (one year or less) of myocardial infarction.
4. Patients with any unstable or life-threatening cardiac arrhythmia.
5. Patients who have been hospitalized for heart failure within the past 3 years.
6. Patients with a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed.
7. Patients with known symptomatic prostatic hyperplasia or bladder neck obstruction as defined in exclusion criteria No. 1.
8. Patients with known narrow-angle glaucoma.
9. Patients with asthma or a history of asthma.
10. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis.
11. Patients with known active tuberculosis.
12. Patients with a history of and/or active significant alcohol or drug abuse. See exclusion criterion No. 1.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2080 (Actual)
Dates: Start 2007-09-06 (Actual); Primary Completion 2009-05-05 (Actual); Study Completion 2009-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (178):
- United States (56):
  - 1205.14.061 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1205.14.054 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1205.14.042 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 1205.14.017 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1205.14.022 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 1205.14.046 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1205.14.008 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1205.14.047 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1205.14.037 Boehringer Ingelheim Investigational Site, Sepulveda, California
  - 1205.14.041 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1205.14.027 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1205.14.034 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1205.14.050 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1205.14.013 Boehringer Ingelheim Investigational Site, Bay Pines, Florida
  - 1205.14.016 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1205.14.048 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1205.14.043 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 1205.14.040 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1205.14.007 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1205.14.053 Boehringer Ingelheim Investigational Site, Stockbridge, Georgia
  - 1205.14.014 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1205.14.035 Boehringer Ingelheim Investigational Site, Olathe, Kansas
  - 1205.14.057 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1205.14.052 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1205.14.036 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1205.14.019 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 1205.14.018 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 1205.14.032 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1205.14.033 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 1205.14.044 Boehringer Ingelheim Investigational Site, Brick, New Jersey
  - 1205.14.056 Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - 1205.14.058 Boehringer Ingelheim Investigational Site, Summit, New Jersey
  - 1205.14.010 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1205.14.062 Boehringer Ingelheim Investigational Site, Larchmont, New York
  - 1205.14.028 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 1205.14.030 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1205.14.021 Boehringer Ingelheim Investigational Site, New York, New York
  - 1205.14.059 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1205.14.012 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1205.14.031 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1205.14.003 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1205.14.004 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1205.14.005 Boehringer Ingelheim Investigational Site, Johnston, Rhode Island
  - 1205.14.029 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1205.14.055 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1205.14.020 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1205.14.045 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1205.14.025 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1205.14.060 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1205.14.002 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1205.14.023 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1205.14.024 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1205.14.026 Boehringer Ingelheim Investigational Site, Roanoke, Virginia
  - 1205.14.009 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1205.14.039 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1205.14.001 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
- Canada (9):
  - 1205.14.151 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1205.14.144 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1205.14.148 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1205.14.143 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 1205.14.142 Boehringer Ingelheim Investigational Site, Downsview, Ontario
  - 1205.14.150 Boehringer Ingelheim Investigational Site, Grimsby, Ontario
  - 1205.14.149 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1205.14.146 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1205.14.145 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Germany (33):
  - 1205.14.381 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1205.14.164 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.167 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.168 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.172 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.175 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.177 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.178 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.377 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.382 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.387 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.388 Boehringer Ingelheim Investigational Site, Berlin
  - 1205.14.165 Boehringer Ingelheim Investigational Site, Bonn
  - 1205.14.176 Boehringer Ingelheim Investigational Site, Cottbus
  - 1205.14.171 Boehringer Ingelheim Investigational Site, Dortmund
  - 1205.14.379 Boehringer Ingelheim Investigational Site, Geesthacht
  - 1205.14.174 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 1205.14.173 Boehringer Ingelheim Investigational Site, Hamburg
  - 1205.14.375 Boehringer Ingelheim Investigational Site, Hanover
  - 1205.14.378 Boehringer Ingelheim Investigational Site, Koblenz
  - 1205.14.170 Boehringer Ingelheim Investigational Site, Lübeck
  - 1205.14.162 Boehringer Ingelheim Investigational Site, Mainz
  - 1205.14.384 Boehringer Ingelheim Investigational Site, Marburg
  - 1205.14.166 Boehringer Ingelheim Investigational Site, Minden
  - 1205.14.372 Boehringer Ingelheim Investigational Site, Neumünster
  - 1205.14.386 Boehringer Ingelheim Investigational Site, Neuruppin
  - 1205.14.385 Boehringer Ingelheim Investigational Site, Oschersleben
  - 1205.14.169 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1205.14.179 Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - 1205.14.376 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 1205.14.374 Boehringer Ingelheim Investigational Site, Schwetzingen
  - 1205.14.371 Boehringer Ingelheim Investigational Site, Witten
  - 1205.14.373 Boehringer Ingelheim Investigational Site, Witten
- Hungary (19):
  - 1205.14.279 Boehringer Ingelheim Investigational Site, Budakeszi
  - 1205.14.273 Boehringer Ingelheim Investigational Site, Budapest
  - 1205.14.283 Boehringer Ingelheim Investigational Site, Budapest
  - 1205.14.287 Boehringer Ingelheim Investigational Site, Budapest
  - 1205.14.286 Boehringer Ingelheim Investigational Site, Cegléd
  - 1205.14.281 Boehringer Ingelheim Investigational Site, Debrecen
  - 1205.14.272 Boehringer Ingelheim Investigational Site, Deszk
  - 1205.14.289 Boehringer Ingelheim Investigational Site, Deszk
  - 1205.14.271 Boehringer Ingelheim Investigational Site, Érd
  - 1205.14.276 Boehringer Ingelheim Investigational Site, Gödöllö
  - 1205.14.282 Boehringer Ingelheim Investigational Site, Gyula
  - 1205.14.277 Boehringer Ingelheim Investigational Site, Komárom
  - 1205.14.278 Boehringer Ingelheim Investigational Site, Mátraháza
  - 1205.14.280 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 1205.14.285 Boehringer Ingelheim Investigational Site, Sopron
  - 1205.14.275 Boehringer Ingelheim Investigational Site, Szarvas
  - 1205.14.288 Boehringer Ingelheim Investigational Site, Százhalombatta
  - 1205.14.284 Boehringer Ingelheim Investigational Site, Tatabánya
  - 1205.14.274 Boehringer Ingelheim Investigational Site, Zalaegerszeg
- Mexico (8):
  - 1205.14.108 Boehringer Ingelheim Investigational Site, Cuernavaca, Mor. México
  - 1205.14.101 Boehringer Ingelheim Investigational Site, Hermosillo, Sonora
  - 1205.14.119 Boehringer Ingelheim Investigational Site, Metepec
  - 1205.14.117 Boehringer Ingelheim Investigational Site, Mexico City
  - 1205.14.120 Boehringer Ingelheim Investigational Site, Mexico City
  - 1205.14.102 Boehringer Ingelheim Investigational Site, Monterrey
  - 1205.14.116 Boehringer Ingelheim Investigational Site, Monterrey, Nuevo León
  - 1205.14.105 Boehringer Ingelheim Investigational Site, Zapopan, Jal.
- Poland (14):
  - 1205.14.251 Boehringer Ingelheim Investigational Site, Chrzanów
  - 1205.14.253 Boehringer Ingelheim Investigational Site, Gdansk
  - 1205.14.254 Boehringer Ingelheim Investigational Site, Gdansk
  - 1205.14.246 Boehringer Ingelheim Investigational Site, Krakow
  - 1205.14.241 Boehringer Ingelheim Investigational Site, Lodz
  - 1205.14.242 Boehringer Ingelheim Investigational Site, Lodz
  - 1205.14.255 Boehringer Ingelheim Investigational Site, Miechów
  - 1205.14.248 Boehringer Ingelheim Investigational Site, Ruda Śląska
  - 1205.14.249 Boehringer Ingelheim Investigational Site, Tarnowskie Góry
  - 1205.14.252 Boehringer Ingelheim Investigational Site, Wilkowice
  - 1205.14.243 Boehringer Ingelheim Investigational Site, Wroclaw
  - 1205.14.244 Boehringer Ingelheim Investigational Site, Wroclaw
  - 1205.14.245 Boehringer Ingelheim Investigational Site, Wroclaw
  - 1205.14.247 Boehringer Ingelheim Investigational Site, Zabrze
- Russia (14):
  - 1205.14.301 Boehringer Ingelheim Investigational Site, Moscow
  - 1205.14.302 Boehringer Ingelheim Investigational Site, Moscow
  - 1205.14.303 Boehringer Ingelheim Investigational Site, Moscow
  - 1205.14.304 Boehringer Ingelheim Investigational Site, Moscow
  - 1205.14.305 Boehringer Ingelheim Investigational Site, Moscow
  - 1205.14.306 Boehringer Ingelheim Investigational Site, Moscow
  - 1205.14.310 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1205.14.311 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1205.14.312 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1205.14.313 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1205.14.314 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1205.14.307 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1205.14.308 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1205.14.309 Boehringer Ingelheim Investigational Site, Yaroslavl
- South Korea (8):
  - 1205.14.225 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 1205.14.228 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 1205.14.227 Boehringer Ingelheim Investigational Site, Seongdong-gu
  - 1205.14.221 Boehringer Ingelheim Investigational Site, Seoul
  - 1205.14.222 Boehringer Ingelheim Investigational Site, Seoul
  - 1205.14.223 Boehringer Ingelheim Investigational Site, Seoul
  - 1205.14.224 Boehringer Ingelheim Investigational Site, Seoul
  - 1205.14.226 Boehringer Ingelheim Investigational Site, Seoul
- Spain (8):
  - 1205.14.182 Boehringer Ingelheim Investigational Site, Badajoz
  - 1205.14.186 Boehringer Ingelheim Investigational Site, Cáceres
  - 1205.14.183 Boehringer Ingelheim Investigational Site, Madrid
  - 1205.14.191 Boehringer Ingelheim Investigational Site, Málaga
  - 1205.14.181 Boehringer Ingelheim Investigational Site, Terrassa (Barcelona)
  - 1205.14.190 Boehringer Ingelheim Investigational Site, Torrevieja
  - 1205.14.189 Boehringer Ingelheim Investigational Site, Valencia
  - 1205.14.187 Boehringer Ingelheim Investigational Site, Vigo
- Taiwan (9):
  - 1205.14.207 Boehringer Ingelheim Investigational Site, Changhua
  - 1205.14.208 Boehringer Ingelheim Investigational Site, Chiayi City
  - 1205.14.210 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1205.14.209 Boehringer Ingelheim Investigational Site, Kaohsiung County
  - 1205.14.205 Boehringer Ingelheim Investigational Site, Taichung
  - 1205.14.206 Boehringer Ingelheim Investigational Site, Taichung
  - 1205.14.202 Boehringer Ingelheim Investigational Site, Taipei
  - 1205.14.204 Boehringer Ingelheim Investigational Site, Taipei
  - 1205.14.201 Boehringer Ingelheim Investigational Site, Taoyuan

REFERENCES:
- [Derived] Abrahams R, Moroni-Zentgraf P, Ramsdell J, Schmidt H, Joseph E, Karpel J. Safety and efficacy of the once-daily anticholinergic BEA2180 compared with tiotropium in patients with COPD. Respir Med. 2013 Jun;107(6):854-62. doi: 10.1016/j.rmed.2013.02.005. Epub 2013 Mar 13. PMID 23490224
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multinational, randomized, double-blind, placebo-and active-controlled, parallel group efficacy and safety comparison of BEA 2180 to tiotropium and placebo delivered by the Respimat® inhaler in patients with chronic obstructive pulmonary disease (COPD).
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects visited specialist site to ensure that they met all implemented inclusion criteria. Subjects meeting the exclusion criteria were excluded.
Groups:
- Placebo: Oral inhalation of solution of Placebo matching BEA 2180 BR was administered once daily via Respimat® inhaler for 24 weeks.
- BEA 2180 BR 50 Microgram (mcg): 2 oral inhalations of solution of 25 micrograms (mcg) of BEA 2180 BR (total: 50 mcg) were administered via Respimat® inhaler once daily for 24 weeks.
- BEA 2180 BR 100 Microgram (mcg): 2 oral inhalations of solution of 50 micrograms (mcg) of BEA 2180 BR (total: 100 mcg) were administered via Respimat® inhaler once daily for 24 weeks.
- BEA 2180 BR 200 Microgram (mcg): 2 oral inhalations of solution of 100 micrograms (mcg) of BEA 2180 BR (total: 200 mcg) were administered via Respimat® inhaler once daily for 24 weeks.
- Tiotropium Bromide 5 Microgram (mcg): 2 inhalation of solution of 2.5 micrograms (mcg) of Tiotropium Bromide (total: 5 mcg) were administered orally via Respimat® inhaler once daily for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Started | 429 | 419 | 415 | 390 | 427
Completed | 365 | 395 | 372 | 340 | 390
Not Completed | 64 | 24 | 43 | 50 | 37
Not completed — Other reasons than listing | 6 | 7 | 14 | 11 | 5
Not completed — Refused continue medication | 16 | 0 | 3 | 3 | 6
Not completed — Lost to Follow-up | 2 | 0 | 4 | 1 | 3
Not completed — Protocol Violation | 1 | 2 | 3 | 3 | 2
Not completed — Lack of Efficacy | 7 | 2 | 1 | 3 | 3
Not completed — Adverse Event | 32 | 13 | 18 | 29 | 18

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The treated set was defined as all patients who were randomized and who took at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg) | Total
Number analyzed (Participants) | 429 | 419 | 415 | 390 | 427 | 2080
Age, Continuous [Mean (Standard Deviation); unit: Year] | 64.41 (8.57) | 63.98 (8.66) | 64.60 (9.11) | 63.89 (8.88) | 63.91 (8.74) | 64.16 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 152 | 146 | 140 | 146 | 739
  Male | 274 | 267 | 269 | 250 | 281 | 1341
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 6 | 4 | 0 | 14
  Asian | 35 | 34 | 34 | 31 | 34 | 168
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 13 | 12 | 15 | 11 | 58
  White | 384 | 371 | 363 | 340 | 382 | 1840
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: liter] — Baseline FEV1 was pre-treatment FEV1 values measured at Day 1 of treatment period (baseline, Visit 2) prior to administration of the first dose of study medication, which was the mean of the measurements obtaining from the pulmonary function tests taken at 40 and 15 minutes prior to drug administration at Day 1 of treatment period.
  liter | 1.18 (0.46) | 1.18 (0.46) | 1.18 (0.48) | 1.19 (0.49) | 1.20 (0.47) | 1.18 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) Response After 24 Weeks
Description: Trough Forced expiratory volume in one second (FEV1) response was defined as the change from baseline in trough FEV1. Trough FEV1 was defined as the mean of the two FEV1 measurements recorded at the pre-dose measurements (40 and 15 minutes before the drug administration) at the end of the dosing interval (24 hours post previous drug administration from the Respimat® Inhaler). Baseline FEV1 was pre-treatment FEV1 values measured at Day 1 of treatment period (baseline) prior to administration of the first dose of study medication, which was the mean of the measurements recorded from the pulmonary function tests taken at 40 and 15 minutes prior to drug administration at Day 1 of treatment period.
Time Frame: 40 minutes (min) and 15 min before drug administration at baseline (Day 1 of treatment period) and Week 24.
Population: The full analysis set (FAS) was defined as all patients in treated set with at least baseline Forced expiratory volume in one second (FEV1) data and at least one acceptable post-treatment trough FEV1 measurement.
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre | -0.034 (0.010) | 0.044 (0.010) | 0.066 (0.011) | 0.087 (0.011) | 0.092 (0.010)

2. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) Response After 1, 2, 4, 8, 12, and 18 Weeks
Description: as for outcome 1
Time Frame: 40 minutes (min) and 15 min before drug administration at baseline (Day 1 of treatment period) and Week 1, 2, 4, 8, 12 and 18.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Groups:
- BEA 2180 BR Inhalation Solution 50 Microgram (mcg): Inhalation of solution of 50 microgram (mcg) BEA 1280 BR (2 inhalations via Respimat® inhaler x 25 mcg) for oral inhalation once daily for 24 weeks.
- BEA 2180 BR Inhalation Solution 100 Microgram (mcg): Inhalation of solution of 100 microgram (mcg) BEA 1280 BR (2 inhalations viaRespimat® inhaler x 50 mcg) for oral inhalation once daily for 24 weeks.
- BEA 2180 BR Inhalation Solution 200 Microgram (mcg): Inhalation of solution of 200 microgram (mcg) BEA 1280 BR (2 inhalations viaRespimat® inhaler x 100 mcg) for oral inhalation once daily for 24 weeks.
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 1 | -0.014 (0.008) | 0.070 (0.008) | 0.090 (0.008) | 0.106 (0.009) | 0.097 (0.008)
  Week 2 | -0.013 (0.009) | 0.080 (0.009) | 0.094 (0.009) | 0.110 (0.009) | 0.105 (0.008)
  Week 4 | -0.020 (0.009) | 0.066 (0.009) | 0.090 (0.009) | 0.100 (0.009) | 0.099 (0.009)
  Week 8 | -0.006 (0.010) | 0.078 (0.010) | 0.086 (0.010) | 0.101 (0.010) | 0.104 (0.010)
  Week 12 | -0.010 (0.010) | 0.066 (0.010) | 0.083 (0.010) | 0.107 (0.010) | 0.109 (0.010)
  Week 18 | -0.023 (0.010) | 0.063 (0.010) | 0.072 (0.010) | 0.096 (0.010) | 0.096 (0.010)

3. Secondary Outcome: Trough Forced Vital Capacity (FVC) Response After 1, 2, 4, 8, 12, 18, and 24 Weeks
Description: Trough forced vital capacity (FVC) response was defined as the change from baseline in trough FVC. Trough FVC was defined as the mean of the two FVC measurements recorded at the pre-dose measurements (40 and 15 minutes before drug administration) at the end of the dosing interval (24 hours post previous drug administration from the Respimat® Inhaler), which were obtained through spirometry at the same time points as for forced expiratory volume in one second. Baseline FVC was the mean of the two measurements of FVC taken at 40 and 15 minutes before drug administration at Day 1 of treatment period.
Time Frame: 40 minutes (min) and 15 min before drug administration at baseline (Day 1 of treatment period) and Week 1, 2, 4, 8, 12, 18, and 24.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 1 | -0.002 (0.015) | 0.146 (0.015) | 0.172 (0.016) | 0.186 (0.016) | 0.174 (0.015)
  Week 2 | -0.002 (0.016) | 0.166 (0.016) | 0.177 (0.016) | 0.186 (0.017) | 0.188 (0.016)
  Week 4 | -0.022 (0.016) | 0.132 (0.016) | 0.157 (0.016) | 0.156 (0.017) | 0.169 (0.016)
  Week 8 | 0.006 (0.018) | 0.148 (0.018) | 0.166 (0.018) | 0.173 (0.018) | 0.177 (0.018)
  Week 12 | 0.001 (0.018) | 0.121 (0.018) | 0.155 (0.018) | 0.171 (0.018) | 0.178 (0.018)
  Week 18 | -0.023 (0.018) | 0.117 (0.018) | 0.131 (0.018) | 0.153 (0.019) | 0.146 (0.018)
  Week 24 | -0.044 (0.019) | 0.081 (0.019) | 0.104 (0.019) | 0.132 (0.020) | 0.146 (0.019)

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve From 0 to 3 Hours (AUC0-3h) Response After 0, 4, 12 and 24 Weeks
Description: Forced expiratory volume in one second (FEV1) area under the curve from 0 to 3 hours (AUC0-3h) response after 0, 4, 12 and 24 weeks are reported. The FEV1 AUC0-3h response is the area under the curve from 0 to 3 hours post drug administration for change from baseline values of FEV1. The area under the curve (AUC) is calculated as the area under the curve from 0 to 3 hours at weeks 0, 4, 12 and 24 using the trapezoidal rule and using planned time, divided by the full duration (3 hours) to report in litres. The mean of the pre-dose values (at 40 minutes and 15 minutes before dosing) are used with a time value of zero for calculating the AUC values starting at zero. The baseline FEV1 is the mean of the two measurements taken at 40 and 15 minutes before drug administration at Day 1 of treatment period.
Time Frame: 40 minutes (min) and 15 min before drug administration and 15 min, 30 min, 60 min, 2 hours, 3 hours after drug administration at Week 0 (Day 1 of treatment period), 4, 12, 24.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 0 | 0.029 (0.007) | 0.172 (0.007) | 0.186 (0.007) | 0.177 (0.007) | 0.165 (0.007)
  Week 4 | 0.021 (0.010) | 0.166 (0.010) | 0.175 (0.010) | 0.165 (0.011) | 0.203 (0.010)
  Week 12 | 0.019 (0.011) | 0.164 (0.011) | 0.166 (0.011) | 0.166 (0.011) | 0.203 (0.011)
  Week 24 | -0.007 (0.011) | 0.140 (0.011) | 0.150 (0.011) | 0.146 (0.012) | 0.177 (0.011)

5. Secondary Outcome: Forced Vital Capacity (FVC) Area Under the Curve From 0 to 3 Hours (AUC0-3h) Response After 0, 4, 12 and 24 Weeks
Description: Forced vital capacity (FVC) area under the curve from 0 to 3 hours (AUC0-3h) response after 0, 4, 12 and 24 weeks are reported. The FVC AUC0-3h response is the area under the curve from 0 to 3 hours post drug administration for change from baseline values of FVC. The area under the curve (AUC) is calculated as the area under the curve from 0 to 3 hours at weeks 0, 4, 12 and 24 using the trapezoidal rule and using planned time, divided by the full duration (3 hours) to report in litres. The mean of the pre-dose values (at 40 minutes and 15 minutes before dosing) are used with a time value of zero for calculating the AUC values starting at zero. The baseline FVC is the mean of the two measurements taken at 40 and 15 minutes before drug administration at Day 1 of treatment period.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 0 | 0.067 (0.015) | 0.321 (0.015) | 0.336 (0.015) | 0.302 (0.015) | 0.312 (0.015)
  Week 4 | 0.050 (0.019) | 0.292 (0.019) | 0.298 (0.020) | 0.247 (0.020) | 0.340 (0.019)
  Week 12 | 0.053 (0.020) | 0.276 (0.020) | 0.278 (0.021) | 0.251 (0.021) | 0.326 (0.020)
  Week 24 | -0.002 (0.021) | 0.233 (0.021) | 0.218 (0.022) | 0.210 (0.022) | 0.274 (0.021)

6. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Peak Response After 0, 4, 12, and 24 Weeks
Description: Forced expiratory volume in one second (FEV1) peak response after 0, 4, 12, and 24 weeks were reported. Peak FEV1 response was the maximum change from baseline for the post-dose measurements of FEV1. Baseline FEV1 is the mean of the two measurements taken at 40 and 15 minutes before drug administration.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 0 | 0.103 (0.008) | 0.246 (0.008) | 0.260 (0.08) | 0.266 (0.009) | 0.246 (0.008)
  Week 4 | 0.090 (0.011) | 0.237 (0.011) | 0.250 (0.011) | 0.243 (0.011) | 0.274 (0.011)
  Week 12 | 0.078 (0.011) | 0.236 (0.011) | 0.236 (0.012) | 0.241 (0.012) | 0.273 (0.011)
  Week 24 | 0.051 (0.012) | 0.207 (0.012) | 0.216 (0.012) | 0.216 (0.012) | 0.242 (0.012)

7. Secondary Outcome: Forced Vital Capacity (FVC) Peak Response After 0, 4, 12, and 24 Weeks
Description: Forced Vital Capacity (FVC) peak response after 0, 4, 12, and 24 weeks were reported. Peak FVC response was the maximum change from baseline for the post-dose measurements of FVC. Baseline FVC is the mean of the two measurements taken at 40 and 15 minutes before drug administration.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 0 | 0.216 (0.018) | 0.474 (0.018) | 0.478 (0.018) | 0.463 (0.019) | 0.463 (0.018)
  Week 4 | 0.186 (0.021) | 0.434 (0.021) | 0.449 (0.021) | 0.386 (0.022) | 0.479 (0.021)
  Week 12 | 0.177 (0.022) | 0.417 (0.022) | 0.412 (0.023) | 0.384 (0.023) | 0.463 (0.022)
  Week 24 | 0.122 (0.023) | 0.369 (0.023) | 0.345 (0.023) | 0.335 (0.024) | 0.393 (0.023)

8. Secondary Outcome: Individual Forced Expiratory Volume in One Second (FEV1) Measurements at Each Time Point
Description: Individual Forced expiratory volume in one second (FEV1) values measured at each time points at Week 0, 4, 12, and 24 were reported.
Time Frame: 15 minutes (min), 30 min, 1 hour (h), 2 h, 3 h after drug administration at Week 0 (Day 1 of treatment period), 4, 12, and 24. At 0 min (at drug administration) at Week 4, 12, and 24.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 0 - 15 minutes (min) | 1.200 (0.006) | 1.309 (0.006) | 1.310 (0.006) | 1.263 (0.006) | 1.276 (0.006)
  Week 0 - 30 min | 1.206 (0.007) | 1.347 (0.007) | 1.357 (0.007) | 1.318 (0.007) | 1.311 (0.007)
  Week 0 - 1 hour (h) | 1.223 (0.008) | 1.375 (0.008) | 1.390 (0.008) | 1.369 (0.008) | 1.353 (0.008)
  Week 0 - 2 h | 1.212 (0.008) | 1.373 (0.008) | 1.388 (0.008) | 1.395 (0.008) | 1.378 (0.008)
  Week 0 - 3 h | 1.220 (0.009) | 1.363 (0.009) | 1.389 (0.009) | 1.403 (0.009) | 1.388 (0.009)
  Week 4 - 0 min | 1.163 (0.009) | 1.249 (0.009) | 1.274 (0.009) | 1.284 (0.009) | 1.283 (0.009)
  Week 4 - 15 min | 1.187 (0.010) | 1.319 (0.010) | 1.321 (0.010) | 1.279 (0.010) | 1.348 (0.010)
  Week 4 - 30 min | 1.200 (0.010) | 1.346 (0.010) | 1.346 (0.011) | 1.308 (0.011) | 1.374 (0.010)
  Week 4 - 1 h | 1.207 (0.011) | 1.360 (0.011) | 1.366 (0.011) | 1.350 (0.011) | 1.397 (0.011)
  Week 4 - 2 h | 1.211 (0.011) | 1.360 (0.011) | 1.372 (0.011) | 1.372 (0.011) | 1.401 (0.011)
  Week 4 - 3 h | 1.211 (0.011) | 1.355 (0.011) | 1.368 (0.011) | 1.380 (0.012) | 1.401 (0.011)
  Week 12 - 0 min | 1.174 (0.010) | 1.249 (0.010) | 1.267 (0.010) | 1.291 (0.010) | 1.293 (0.010)
  Week 12 - 15 min | 1.188 (0.011) | 1.321 (0.011) | 1.313 (0.011) | 1.292 (0.011) | 1.354 (0.011)
  Week 12 - 30 min | 1.196 (0.011) | 1.348 (0.011) | 1.335 (0.011) | 1.313 (0.011) | 1.371 (0.011)
  Week 12 - 1 h | 1.209 (0.011) | 1.358 (0.011) | 1.356 (0.011) | 1.345 (0.011) | 1.391 (0.011)
  Week 12 - 2 h | 1.205 (0.011) | 1.357 (0.011) | 1.365 (0.011) | 1.372 (0.012) | 1.401 (0.011)
  Week 12 - 3 h | 1.205 (0.011) | 1.352 (0.012) | 1.363 (0.012) | 1.384 (0.012) | 1.401 (0.011)
  Week 24 - 0 min | 1.150 (0.010) | 1.227 (0.010) | 1.250 (0.011) | 1.270 (0.011) | 1.276 (0.010)
  Week 24 0:15 min | 1.164 (0.011) | 1.297 (0.011) | 1.298 (0.011) | 1.278 (0.012) | 1.326 (0.011)
  Week 24 - 30 min | 1.170 (0.011) | 1.318 (0.012) | 1.320 (0.012) | 1.296 (0.012) | 1.355 (0.011)
  Week 24 - 1 h | 1.180 (0.012) | 1.338 (0.012) | 1.342 (0.012) | 1.331 (0.012) | 1.368 (0.012)
  Week 24 - 2 h | 1.180 (0.012) | 1.332 (0.012) | 1.345 (0.012) | 1.346 (0.012) | 1.373 (0.012)
  Week 24 - 3 h | 1.180 (0.012) | 1.326 (0.012) | 1.344 (0.012) | 1.357 (0.012) | 1.370 (0.012)

9. Secondary Outcome: Individual Forced Vital Capacity (FVC) Measurements at Each Time Point
Description: Individual Forced Vital Capacity (FVC) values measured at each time point at Week 0, 4, 12, and 24 were reported.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litre
  Week 0 - 15 minutes (min) | 2.572 (0.013) | 2.787 (0.013) | 2.778 (0.013) | 2.691 (0.013) | 2.729 (0.013)
  Week 0 - 30 min | 2.589 (0.015) | 2.854 (0.015) | 2.852 (0.015) | 2.776 (0.016) | 2.802 (0.015)
  Week 0 - 1 hour (h) | 2.617 (0.016) | 2.885 (0.017) | 2.907 (0.017) | 2.853 (0.017) | 2.864 (0.016)
  Week 0 - 2 h | 2.598 (0.017) | 2.881 (0.017) | 2.896 (0.018) | 2.886 (0.018) | 2.885 (0.017)
  Week 0 - 3 h | 2.617 (0.019) | 2.867 (0.019) | 2.896 (0.019) | 2.896 (0.019) | 2.901 (0.019)
  Week 4 - 0 minutes | 2.510 (0.016) | 2.665 (0.016) | 2.689 (0.016) | 2.688 (0.017) | 2.702 (0.016)
  Week 4 - 15 minutes | 2.547 (0.019) | 2.770 (0.019) | 2.776 (0.019) | 2.670 (0.019) | 2.822 (0.019)
  Week 4 - 30 min | 2.575 (0.020) | 2.812 (0.020) | 2.803 (0.020) | 2.711 (0.020) | 2.852 (0.020)
  Week 4 - 1 h | 2.590 (0.020) | 2.842 (0.020) | 2.848 (0.021) | 2.779 (0.021) | 2.891 (0.020)
  Week 4 - 2 h | 2.592 (0.021) | 2.842 (0.021) | 2.851 (0.021) | 2.815 (0.022) | 2.893 (0.021)
  Week 4 - 3 h | 2.595 (0.021) | 2.842 (0.021) | 2.849 (0.022) | 2.837 (0.022) | 2.891 (0.021)
  Week 12 - 0 min | 2.533 (0.018) | 2.654 (0.018) | 2.687 (0.018) | 2.703 (0.018) | 2.711 (0.018)
  Week 12 - 15 min | 2.563 (0.020) | 2.764 (0.020) | 2.751 (0.020) | 2.688 (0.021) | 2.803 (0.020)
  Week 12 - 30 minutes | 2.574 (0.020) | 2.796 (0.020) | 2.788 (0.021) | 2.720 (0.021) | 2.844 (0.020)
  Week 12 - 1 h | 2.606 (0.021) | 2.823 (0.021) | 2.821 (0.022) | 2.773 (0.022) | 2.866 (0.021)
  Week 12 - 2 h | 2.584 (0.022) | 2.828 (0.022) | 2.829 (0.022) | 2.820 (0.023) | 2.878 (0.022)
  Week 12 - 3 h | 2.588 (0.022) | 2.819 (0.022) | 2.836 (0.022) | 2.840 (0.023) | 2.886 (0.022)
  Week 24 - 0 min | 2.489 (0.019) | 2.614 (0.019) | 2.637 (0.019) | 2.664 (0.020) | 2.678 (0.019)
  Week 24 - 15 min | 2.504 (0.021) | 2.725 (0.021) | 2.705 (0.021) | 2.667 (0.022) | 2.761 (0.021)
  Week 24- 30 min | 2.520 (0.022) | 2.753 (0.022) | 2.724 (0.022) | 2.690 (0.022) | 2.803 (0.022)
  Week 24 - 1 h | 2.539 (0.022) | 2.793 (0.022) | 2.763 (0.022) | 2.739 (0.023) | 2.823 (0.022)
  Week 24 - 2 h | 2.533 (0.023) | 2.778 (0.023) | 2.770 (0.023) | 2.771 (0.023) | 2.822 (0.022)
  Week 24 - 3 h | 2.547 (0.023) | 2.769 (0.024) | 2.766 (0.024) | 2.789 (0.024) | 2.806 (0.023)

10. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) Response on Day 3 and 5
Description: Trough Forced expiratory volume in one second (FEV1) response on Day 3 and 5 are reported, for which the FEV1 response is the change from baseline in trough FEV1. Trough FEV1 for respective day (Day 3 or Day 5)was defined as the mean of the two FEV1 measurements recorded at the pre-dose measurements (40 and 15 minutes before the drug administration) at the end of the dosing interval (24 hours post previous drug administration from the Respimat® Inhaler) at that day. Baseline FEV1 was pre-treatment FEV1 values measured at Day 1 of treatment period (baseline) prior to administration of the first dose of study medication, which was the mean of the measurements recorded from the pulmonary function tests taken at 40 and 15 minutes prior to drug administration at Day 1 of treatment period.
Time Frame: 40 minutes (min) and 15 min before drug administration at Day 1 (baseline) and Day 3 and 5 of treatment period.
Population: Sub-study set (SUB): This patient set includes all patients in the full analysis set that were enrolled in the sub-study (at selected sites only) and have acceptable non-missing forced expiratory volume in one second (FEV1) data from 2 additional visits on Day 3 and 5.
Measure: Mean (Standard Error); unit: liter
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 55 | 58 | 56 | 54 | 53
liter
  Day 3 | 0.008 (0.026) | 0.060 (0.025) | 0.101 (0.025) | 0.124 (0.026) | 0.103 (0.026)
  Day 5 | 0.012 (0.023) | 0.041 (0.023) | 0.095 (0.023) | 0.115 (0.24) | 0.118 (0.024)

11. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) at 3 Minutes and 10 Minutes Following Drug Administration
Description: Forced expiratory volume in one second (FEV1) values at 3 minutes and 10 minutes following drug administration at Week 0, 4, 12, and 24 are reported.
Time Frame: 3 minutes (min) and 10 after drug administration at Week 0 (Day 1 of treatment period), 4, 12, and 24.
Population: as for outcome 10
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 55 | 58 | 56 | 54 | 53
litre
  Week 0 - 3 minutes (min) | 1.128 (0.015) | 1.195 (0.015) | 1.185 (0.015) | 1.147 (0.015) | 1.206 (0.016)
  Week 0 -10 min | 1.135 (0.018) | 1.253 (0.017) | 1.268 (0.017) | 1.224 (0.018) | 1.247 (0.018)
  Week 4 - 3 min | 1.161 (0.026) | 1.208 (0.025) | 1.259 (0.025) | 1.227 (0.026) | 1.260 (0.026)
  Week 4 - 10 min | 1.160 (0.028) | 1.252 (0.027) | 1.312 (0.028) | 1.252 (0.028) | 1.301 (0.029)
  Week 12 - 3 min | 1.151 (0.028) | 1.233 (0.027) | 1.251 (0.027) | 1.258 (0.028) | 1.310 (0.028)
  Week 12 - 10 min | 1.172 (0.027) | 1.258 (0.027) | 1.304 (0.027) | 1.279 (0.027) | 1.336 (0.028)
  Week 24 - 3 min | 1.115 (0.029) | 1.196 (0.029) | 1.230 (0.029) | 1.211 (0.030) | 1.301 (0.030)
  Week 24 - 10 min | 1.138 (0.032) | 1.240 (0.031) | 1.278 (0.031) | 1.244 (0.032) | 1.329 (0.032)

12. Secondary Outcome: Forced Vital Capacity (FVC) at 3 Minutes and 10 Minutes Following Drug Administration
Description: Forced Vital Capacity (FVC) values at 3 minutes and 10 minutes following drug administration at Week 0, 4, 12, and 24 are reported.
Time Frame: 3 minutes (min) and 10 min after drug administration at Week 0 (Day 1 of treatment period), 4, 12, and 24.
Population: as for outcome 10
Measure: Mean (Standard Error); unit: litre
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 55 | 58 | 56 | 54 | 53
litre
  Week 0 - 3 minutes (min) | 2.381 (0.028) | 2.530 (0.027) | 2.535 (0.027) | 2.455 (0.028) | 2.500 (0.028)
  Week 0 - 10 min | 2.392 (0.034) | 2.624 (0.033) | 2.658 (0.033) | 2.557 (0.034) | 2.593 (0.034)
  Week 4 - 3 min | 2.391 (0.044) | 2.623 (0.043) | 2.638 (0.044) | 2.523 (0.044) | 2.601 (0.045)
  Week 4 - 10 min | 2.391 (0.049) | 2.693 (0.048) | 2.697 (0.048) | 2.540 (0.049) | 2.634 (0.050)
  Week 12 - 3 min | 2.395 (0.048) | 2.594 (0.047) | 2.604 (0.048) | 2.549 (0.049) | 2.631 (0.049)
  Week 12 - 10 min | 2.417 (0.050) | 2.648 (0.049) | 2.637 (0.049) | 2.579 (0.050) | 2.646 (0.051)
  Week 24 - 3 min | 2.355 (0.054) | 2.566 (0.053) | 2.556 (0.053) | 2.513 (0.054) | 2.624 (0.055)
  Week 24 - 10 min | 2.403 (0.058) | 2.635 (0.057) | 2.599 (0.057) | 2.545 (0.058) | 2.664 (0.059)

13. Secondary Outcome: Weekly Mean Pre-dose Morning Peak Expiratory Flow Rate (PEFR)
Description: The patient recorded twice daily peak flow measurements with an electronic peak flow meter throughout the entire evaluation period. Morning measurements were performed immediately upon arising after the patient had cleared out mucus, prior to administration of trial and/or rescue medication. The evening measurements were performed at bedtime. The weekly mean morning peak expiratory flow rate (PEFR) is reported.
Time Frame: Assessed before drug administration per day during 24 weeks with weekly mean values reporting.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litres/minute
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litres/minute
  Week 1 | 163.41 (1.629) | 177.03 (1.641) | 176.20 (1.658) | 179.46 (1.718) | 177.54 (1.628)
  Week 2 | 164.34 (1.917) | 177.64 (1.932) | 175.82 (1.952) | 179.24 (2.023) | 176.46 (1.916)
  Week 3 | 164.53 (1.957) | 177.19 (1.972) | 177.38 (1.993) | 178.94 (2.067) | 175.49 (1.956)
  Week 4 | 163.82 (2.006) | 174.99 (2.021) | 176.37 (2.042) | 178.06 (2.118) | 175.17 (2.004)
  Week 5 | 163.00 (1.983) | 176.16 (1.998) | 176.90 (2.019) | 178.29 (2.094) | 176.32 (1.982)
  Week 6 | 162.31 (2.058) | 176.26 (2.073) | 175.31 (2.095) | 177.59 (2.172) | 175.09 (2.056)
  Week 7 | 160.30 (2.033) | 175.71 (2.049) | 174.35 (2.070) | 175.85 (2.147) | 175.50 (2.032)
  Week 8 | 159.83 (2.085) | 173.99 (2.101) | 173.95 (2.123) | 176.41 (2.201) | 174.71 (2.084)
  Week 9 | 159.89 (2.156) | 175.74 (2.171) | 172.84 (2.194) | 177.35 (2.274) | 174.75 (2.154)
  Week 10 | 158.74 (2.126) | 173.63 (2.142) | 171.24 (2.164) | 176.14 (2.242) | 174.71 (2.125)
  Week 11 | 157.98 (2.165) | 173.45 (2.181) | 169.92 (2.204) | 174.05 (2.283) | 174.82 (2.163)
  Week 12 | 156.91 (2.192) | 174.72 (2.209) | 169.90 (2.232) | 175.40 (2.316) | 174.63 (2.191)
  Week 13 | 156.22 (2.093) | 173.59 (2.109) | 169.96 (2.131) | 175.51 (2.211) | 175.97 (2.091)
  Week 14 | 156.66 (2.165) | 172.29 (2.181) | 168.51 (2.203) | 175.65 (2.283) | 174.86 (2.163)
  Week 15 | 156.78 (2.196) | 171.12 (2.213) | 168.69 (2.236) | 175.01 (2.318) | 174.03 (2.195)
  Week 16 | 155.76 (2.206) | 170.92 (2.223) | 169.26 (2.246) | 174.07 (2.330) | 174.23 (2.205)
  Week 17 | 154.59 (2.267) | 171.32 (2.285) | 169.53 (2.309) | 174.89 (2.396) | 174.04 (2.266)
  Week 18 | 154.04 (2.248) | 169.36 (2.266) | 168.95 (2.289) | 173.59 (2.376) | 171.90 (2.246)
  Week 19 | 154.37 (2.263) | 169.24 (2.280) | 170.45 (2.304) | 175.29 (2.389) | 172.92 (2.261)
  Week 20 | 154.77 (2.291) | 169.31 (2.309) | 169.84 (2.332) | 174.81 (2.420) | 173.31 (2.289)
  Week 21 | 153.47 (2.276) | 169.30 (2.293) | 169.12 (2.317) | 175.43 (2.404) | 172.77 (2.274)
  Week 22 | 153.85 (2.267) | 167.60 (2.284) | 169.29 (2.308) | 175.12 (2.393) | 171.93 (2.265)
  Week 23 | 153.41 (2.303) | 167.38 (2.320) | 167.26 (2.345) | 174.30 (2.430) | 171.13 (2.302)
  Week 24 | 153.15 (2.311) | 167.08 (2.329) | 165.87 (2.353) | 176.36 (2.441) | 171.53 (2.310)

14. Secondary Outcome: Weekly Mean Evening Peak Expiratory Flow Rate (PEFR)
Description: The patient recorded twice daily peak flow measurements with an electronic peak flow meter throughout the entire evaluation period. Morning measurements were performed immediately upon arising after the patient had cleared out mucus, prior to administration of trial and/or rescue medication. The evening measurements were performed at bedtime. The weekly mean of evening peak expiratory flow rate (PEFR) is reported.
Time Frame: Assessed at bed time per day during 24 weeks with weekly mean values reporting.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litres/minute
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
litres/minute
  Week 1 | 173.64 (1.467) | 186.40 (1.463) | 186.37 (1.467) | 187.31 (1.542) | 187.13 (1.446)
  Week 2 | 173.18 (1.694) | 187.16 (1.690) | 185.96 (1.694) | 187.16 (1.782) | 185.79 (1.669)
  Week 3 | 171.85 (1.761) | 187.14 (1.756) | 183.77 (1.761) | 187.41 (1.851) | 185.61 (1.735)
  Week 4 | 170.91 (1.858) | 186.96 (1.853) | 184.33 (1.858) | 187.11 (1.952) | 185.23 (1.831)
  Week 5 | 172.33 (1.921) | 186.03 (1.915) | 186.84 (1.920) | 185.67 (2.017) | 185.02 (1.893)
  Week 6 | 169.29 (2.009) | 183.97 (2.004) | 185.32 (2.009) | 184.51 (2.110) | 184.34 (1.980)
  Week 7 | 168.10 (1.989) | 183.82 (1.984) | 184.57 (1.989) | 182.39 (2.090) | 183.80 (1.960)
  Week 8 | 166.98 (1.975) | 183.69 (1.970) | 182.81 (1.975) | 182.01 (2.076) | 181.66 (1.947)
  Week 9 | 165.67 (2.033) | 182.98 (2.028) | 181.88 (2.033) | 184.21 (2.136) | 183.38 (2.004)
  Week 10 | 164.15 (2.067) | 181.90 (2.062) | 179.46 (2.067) | 182.53 (2.170) | 182.12 (2.038)
  Week 11 | 163.02 (2.122) | 182.05 (2.117) | 179.36 (2.122) | 182.54 (2.227) | 181.58 (2.092)
  Week 12 | 163.84 (2.169) | 180.46 (2.163) | 179.65 (2.169) | 180.52 (2.281) | 181.09 (2.138)
  Week 13 | 163.95 (2.162) | 180.80 (2.156) | 178.40 (2.162) | 181.12 (2.270) | 183.50 (2.131)
  Week 14 | 162.72 (2.168) | 179.23 (2.162) | 177.70 (2.168) | 181.26 (2.278) | 183.27 (2.137)
  Week 15 | 162.77 (2.193) | 178.86 (2.187) | 177.33 (2.193) | 181.66 (2.304) | 182.12 (2.162)
  Week 16 | 161.50 (2.227) | 179.17 (2.220) | 177.30 (2.226) | 180.18 (2.342) | 180.76 (2.194)
  Week 17 | 161.12 (2.199) | 179.50 (2.193) | 177.51 (2.198) | 178.95 (2.314) | 180.40 (2.167)
  Week 18 | 161.66 (2.206) | 177.88 (2.200) | 176.28 (2.206) | 178.92 (2.321) | 179.47 (2.174)
  Week 19 | 161.70 (2.229) | 177.34 (2.223) | 177.78 (2.229) | 178.64 (2.342) | 179.98 (2.197)
  Week 20 | 160.54 (2.322) | 177.50 (2.316) | 177.23 (2.322) | 179.20 (2.441) | 180.70 (2.288)
  Week 21 | 161.13 (2.307) | 175.87 (2.300) | 176.16 (2.306) | 178.87 (2.424) | 179.66 (2.273)
  Week 22 | 160.32 (2.309) | 174.78 (2.302) | 175.23 (2.308) | 177.71 (2.424) | 178.98 (2.275)
  Week 23 | 160.75 (2.316) | 174.37 (2.310) | 176.10 (2.316) | 177.54 (2.434) | 178.20 (2.283)
  Week 24 | 159.69 (2.356) | 172.72 (2.349) | 176.20 (2.356) | 179.04 (2.475) | 178.21 (2.322)

15. Secondary Outcome: Weekly Mean Number of Occasions of Rescue Therapy Used Per Day (as Occasion Requires (PRN) Salbutamol [Albuterol])
Description: The patient recorded the number of occasions salbutamol (albuterol) Metered Dose Inhaler (MDI) was used each day and night during the entire evaluation period. The weekly mean number of occasions of rescue therapy used per day (PRN salbutamol [albuterol]) is reported.
Time Frame: Assessed once per day during 24 weeks with weekly mean values reporting.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Metered Dose Inhaler use per day
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
Metered Dose Inhaler use per day
  Week 1 | 2.514 (0.075) | 1.964 (0.075) | 1.972 (0.076) | 1.790 (0.078) | 2.084 (0.075)
  Week 2 | 2.524 (0.079) | 1.985 (0.079) | 2.044 (0.080) | 1.803 (0.082) | 2.109 (0.079)
  Week 3 | 2.509 (0.081) | 1.960 (0.081) | 2.037 (0.081) | 1.835 (0.084) | 2.093 (0.080)
  Week 4 | 2.498 (0.081) | 1.977 (0.081) | 2.017 (0.082) | 1.885 (0.085) | 2.118 (0.081)
  Week 5 | 2.548 (0.086) | 2.040 (0.085) | 2.012 (0.086) | 1.768 (0.089) | 2.106 (0.085)
  Week 6 | 2.629 (0.088) | 2.048 (0.088) | 2.041 (0.088) | 1.789 (0.091) | 2.116 (0.087)
  Week 7 | 2.656 (0.088) | 2.042 (0.088) | 2.039 (0.088) | 1.851 (0.091) | 2.122 (0.087)
  Week 8 | 2.612 (0.089) | 2.007 (0.088) | 2.010 (0.089) | 1.877 (0.092) | 2.129 (0.088)
  Week 9 | 2.617 (0.088) | 2.026 (0.088) | 1.981 (0.089) | 1.834 (0.092) | 2.094 (0.088)
  Week 10 | 2.623 (0.090) | 2.062 (0.090) | 2.013 (0.091) | 1.838 (0.093) | 2.137 (0.089)
  Week 11 | 2.693 (0.092) | 2.136 (0.092) | 2.020 (0.093) | 1.872 (0.096) | 2.154 (0.091)
  Week 12 | 2.678 (0.091) | 2.127 (0.091) | 2.011 (0.092) | 1.899 (0.095) | 2.122 (0.091)
  Week 13 | 2.645 (0.091) | 2.074 (0.091) | 2.108 (0.092) | 1.844 (0.094) | 2.112 (0.090)
  Week 14 | 2.655 (0.091) | 2.131 (0.091) | 2.161 (0.092) | 1.844 (0.095) | 2.063 (0.091)
  Week 15 | 2.712 (0.094) | 2.148 (0.094) | 2.127 (0.095) | 1.859 (0.098) | 2.141 (0.093)
  Week 16 | 2.732 (0.095) | 2.081 (0.095) | 2.090 (0.096) | 1.906 (0.099) | 2.143 (0.094)
  Week 17 | 2.738 (0.096) | 2.060 (0.096) | 2.111 (0.097) | 1.899 (0.100) | 2.153 (0.096)
  Week 18 | 2.756 (0.097) | 2.074 (0.097) | 2.078 (0.098) | 1.872 (0.100) | 2.146 (0.096)
  Week 19 | 2.706 (0.099) | 2.105 (0.099) | 2.083 (0.100) | 1.896 (0.103) | 2.154 (0.098)
  Week 20 | 2.670 (0.101) | 2.084 (0.101) | 2.149 (0.102) | 1.975 (0.105) | 2.180 (0.100)
  Week 21 | 2.706 (0.098) | 2.103 (0.098) | 2.116 (0.099) | 1.928 (0.102) | 2.156 (0.098)
  Week 22 | 2.704 (0.098) | 2.124 (0.098) | 2.119 (0.099) | 1.928 (0.102) | 2.168 (0.098)
  Week 23 | 2.675 (0.098) | 2.056 (0.098) | 2.094 (0.099) | 1.959 (0.102) | 2.138 (0.097)
  Week 24 | 2.672 (0.100) | 2.114 (0.100) | 2.116 (0.101) | 1.961 (0.104) | 2.148 (0.099)

16. Secondary Outcome: Physician's Global Evaluation
Description: Physicians make a global evaluation reflecting the physician's global opinion of the overall clinical condition of the patient as "poor" (score 1 or 2), "fair" (score 3 or 4), "good" (score 5 or 6), or "excellent" (score 7 or 8). These assessments are made prior to pulmonary function testing and are summarized on pulmonary function test days. This evaluation was based on the need for concomitant medication, number and severity of exacerbations since the last visit, severity of cough, ability to exercise, amount of wheezing, and other relevant clinical observations. The score ranges from 1 to 8 with higher score indicating better overall clinical condition.
Time Frame: At Week 0, 4, 12, and 24.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
Score on scale
  Week 0 | 4.4 (1.2) | 4.5 (1.2) | 4.5 (1.2) | 4.4 (1.2) | 4.5 (1.1)
  Week 4 | 4.541 (0.042) | 4.714 (0.042) | 4.747 (0.042) | 4.807 (0.044) | 4.739 (0.042)
  Week 12 | 4.582 (0.047) | 4.804 (0.047) | 4.790 (0.047) | 4.880 (0.048) | 4.816 (0.047)
  Week 24 | 4.613 (0.053) | 4.865 (0.053) | 4.775 (0.054) | 4.888 (0.055) | 4.810 (0.053)

17. Secondary Outcome: Transition Dyspnea Index - Functional Impairment Domain Score
Description: The transitional dyspnea index (TDI) evaluates the patient's condition related to breathlessness. The TDI includes three domains: functional impairment, magnitude of task, and magnitude of effort. The TDI domain score of functional impairment is reported, which domain score ranges from -3 (major deterioration in the ability of working and doing activities due to shortness of breath; the worst score) to 3 (major improvement in the ability of working and doing activities; mild restriction on full activities due to the improvement of shortness of breath; the best score).
Time Frame: At Week 0 (baseline), 4, 12 and 24.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
Score on a scale
  Week 0 | 2.3 (0.9) | 2.3 (0.9) | 2.3 (0.9) | 2.2 (0.9) | 2.3 (0.9)
  Week 4 | 0.192 (0.048) | 0.379 (0.048) | 0.480 (0.049) | 0.518 (0.050) | 0.462 (0.048)
  Week 12 | 0.276 (0.052) | 0.474 (0.052) | 0.519 (0.053) | 0.454 (0.054) | 0.492 (0.052)
  Week 24 | 0.353 (0.054) | 0.465 (0.054) | 0.445 (0.055) | 0.465 (0.056) | 0.488 (0.054)

18. Secondary Outcome: Transition Dyspnea Index - Magnitude of Task Domain Score
Description: The transitional dyspnea index (TDI) evaluates the patient's condition related to breathlessness. The TDI includes three domains: functional impairment, magnitude of task, and magnitude of effort. The TDI domain score of magnitude of task is reported, which domain score ranges from -3 (major deterioration from baseline status; the worst score) to 3 (major improvement from baseline status; the best score).
Time Frame: At week 0 (baseline), 4, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
Score on a scale
  Week 0 | 2.2 (0.8) | 2.2 (0.8) | 2.2 (0.8) | 2.2 (0.8) | 2.2 (0.7)
  Week 4 | 0.245 (0.048) | 0.494 (0.048) | 0.538 (0.049) | 0.571 (0.050) | 0.489 (0.048)
  Week 12 | 0.282 (0.053) | 0.494 (0.053) | 0.587 (0.053) | 0.479 (0.054) | 0.523 (0.053)
  Week 24 | 0.322 (0.055) | 0.510 (0.055) | 0.513 (0.056) | 0.514 (0.057) | 0.496 (0.055)

19. Secondary Outcome: Transition Dyspnea Index - Magnitude of Effort Domain Score
Description: The transitional dyspnea index (TDI) evaluates the patient's condition related to breathlessness. The TDI includes three domains: functional impairment, magnitude of task, and magnitude of effort. The TDI domain score of magnitude of effort is reported, which sub-score ranges from -3 (severe decrease in effort from baseline to avoid shortness of breath. Activities now take 50-100% longer to complete than required at baseline; the worst score) to 3 (Able to do things with much greater effort than previously with few pauses. Activities may be performed 50- 100% more rapidly than at baseline; the best score).
Time Frame: At Week 0 (baseline), 4, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR Inhalation Solution 50 Microgram (mcg) | BEA 2180 BR Inhalation Solution 100 Microgram (mcg) | BEA 2180 BR Inhalation Solution 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 421 | 417 | 409 | 387 | 423
Score on a scale
  Week 0 | 2.1 (0.7) | 2.0 (0.8) | 2.0 (0.8) | 2.0 (0.7) | 2.0 (0.7)
  Week 4 | 0.161 (0.048) | 0.437 (0.048) | 0.497 (0.049) | 0.478 (0.050) | 0.449 (0.048)
  Week 12 | 0.253 (0.054) | 0.423 (0.054) | 0.486 (0.054) | 0.460 (0.055) | 0.478 (0.053)
  Week 24 | 0.273 (0.057) | 0.458 (0.057) | 0.472 (0.058) | 0.502 (0.059) | 0.474 (0.057)

20. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Total Score
Description: The St. George's Respiratory Questionnaire (SGRQ) is a well-established, self-completed tool measuring health-related quality of life in patients with diseases of airways obstruction on three aspects of symptoms, activity, and impacts. The total SGRQ score is reported, which ranges from 0 (the best score) to 100 (the worst score) with smaller score value indicating less limitations due to breathlessness and better quality of life.
Time Frame: At Week 0, 4, 12, and 24.
Population: The full analysis set (FAS) was defined as all patients in treated set with at least baseline Forced expiratory volume in one second (FEV1) data and at least one acceptable post-treatment trough FEV1 measurement. Only patients with non-missing outcomes are included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 411 | 415 | 404 | 379 | 419
Score on a scale
  Week 0 | 43.2 (18.1) | 41.9 (17.5) | 42.5 (17.7) | 43.8 (18.8) | 43.1 (17.8)
  Week 4 | 41.969 (0.486) | 40.552 (0.484) | 39.865 (0.490) | 40.689 (0.506) | 40.706 (0.481)
  Week 12 | 42.744 (0.575) | 40.293 (0.573) | 39.506 (0.580) | 40.368 (0.596) | 39.489 (0.570)
  Week 24 | 42.993 (0.626) | 40.103 (0.624) | 40.058 (0.632) | 40.728 (0.651) | 39.547 (0.621)

21. Secondary Outcome: 36-item-health Survey (SF-36) 8 Domain Scores at Baseline
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function (10 questions), role physical (4 questions), Bodily pain (2 questions), General physical health (5 questions), Vitality (4 questions), Social functioning (2 questions), role emotional (3 questions), and General mental health (5 questions). Each domain score is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the score value, the better the health condition.
Time Frame: At baseline (Week 0, Day 1 of treatment period).
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Physical function | 50.2 (24.5) | 51.4 (25.1) | 51.9 (24.2) | 49.1 (24.7) | 51.1 (22.9)
  Role physical | 53.9 (27.5) | 55.9 (27.5) | 53.3 (26.7) | 53.9 (27.7) | 54.9 (27.1)
  Bodily pain | 68.9 (26.6) | 68.6 (25.5) | 66.7 (26.7) | 67.1 (26.8) | 65.9 (26.8)
  General physical health | 48.5 (18.5) | 49.2 (18.0) | 48.0 (18.7) | 48.5 (19.2) | 47.1 (18.4)
  Vitality | 53.9 (20.3) | 53.6 (20.1) | 53.4 (21.1) | 52.1 (20.3) | 51.8 (20.3)
  Social functioning | 75.3 (24.0) | 76.2 (22.8) | 75.2 (24.4) | 74.3 (23.9) | 74.2 (23.0)
  Role emotional | 70.0 (28.9) | 70.8 (28.1) | 69.3 (27.6) | 67.8 (29.6) | 68.5 (27.8)
  General mental health | 72.0 (19.2) | 70.4 (19.4) | 71.2 (19.3) | 68.5 (20.0) | 68.5 (19.2)

22. Secondary Outcome: 36-item-health Survey (SF-36) - Physical Function Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of physical function (based on 10 questions) is reported, which is the weighted sum of the questions in corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the better the physical function.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 50.201 (0.726) | 51.831 (0.724) | 52.812 (0.732) | 52.961 (0.754) | 53.052 (0.720)
  Week 12 | 50.541 (0.806) | 52.561 (0.804) | 52.099 (0.813) | 53.716 (0.838) | 53.935 (0.800)
  Week 24 | 50.624 (0.854) | 52.702 (0.851) | 51.631 (0.861) | 52.256 (0.887) | 54.191 (0.847)

23. Secondary Outcome: 36-item-health Survey (SF-36) - Role Physical Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of role limitations due to physical health problems (based on 4 questions) is reported, which is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the less limitations in roles due to physical health problems.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 55.168 (0.962) | 57.326 (0.959) | 57.469 (0.969) | 56.898 (1.000) | 57.950 (0.954)
  Week 12 | 54.405 (0.986) | 57.271 (0.983) | 57.186 (0.993) | 56.938 (1.024) | 57.417 (0.978)
  Week 24 | 53.138 (1.047) | 57.095 (1.044) | 54.934 (1.055) | 55.871 (1.087) | 57.020 (1.038)

24. Secondary Outcome: 36-item-health Survey (SF-36) - Bodily Pain Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of bodily pain (based on 2 questions) is reported, which is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the less severer the bodily pain.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 66.828 (1.024) | 68.184 (1.020) | 70.738 (1.031) | 66.439 (1.063) | 70.512 (1.015)
  Week 12 | 66.749 (1.124) | 66.698 (1.120) | 70.316 (1.132) | 67.815 (1.167) | 70.300 (1.115)
  Week 24 | 64.964 (1.162) | 66.610 (1.158) | 68.279 (1.171) | 66.887 (1.205) | 69.995 (1.153)

25. Secondary Outcome: 36-item-health Survey (SF-36) - General Physical Health Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of general physical health (based on 5 questions) is reported, which is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the better the physical health in general.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 47.187 (0.630) | 48.725 (0.628) | 50.929 (0.635) | 49.476 (0.656) | 50.609 (0.625)
  Week 12 | 46.709 (0.679) | 48.402 (0.677) | 50.057 (0.685) | 49.482 (0.706) | 50.847 (0.674)
  Week 24 | 45.913 (0.718) | 48.520 (0.716) | 50.156 (0.724) | 49.816 (0.746) | 49.477 (0.712)

26. Secondary Outcome: 36-item-health Survey (SF-36) - Vitality Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of vitality (based on 4 questions) is reported, which is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the more vitality and less fatigue one has.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 52.501 (0.716) | 53.516 (0.713) | 54.084 (0.721) | 53.630 (0.743) | 54.881 (0.710)
  Week 12 | 51.676 (0.759) | 53.670 (0.756) | 53.947 (0.765) | 53.935 (0.788) | 55.317 (0.753)
  Week 24 | 51.188 (0.804) | 52.892 (0.801) | 54.080 (0.810) | 54.211 (0.833) | 54.542 (0.798)

27. Secondary Outcome: 36-item-health Survey (SF-36) - Social Functioning Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of Social functioning (based on 2 questions) is reported, which is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the better the social functioning.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 75.574 (0.919) | 76.235 (0.916) | 76.418 (0.926) | 77.177 (0.954) | 77.053 (0.912)
  Week 12 | 73.093 (0.982) | 76.801 (0.979) | 75.108 (0.989) | 75.798 (1.018) | 76.992 (0.974)
  Week 24 | 71.440 (1.062) | 75.157 (1.059) | 74.295 (1.070) | 75.520 (1.102) | 73.993 (1.054)

28. Secondary Outcome: 36-item-health Survey (SF-36) - Role Emotional Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of role emotional (based on 4 questions) is reported, which is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the less limitation in roles due to emotional problems.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 69.365 (1.073) | 70.509 (1.070) | 70.473 (1.081) | 71.646 (1.115) | 71.313 (1.065)
  Week 12 | 67.399 (1.108) | 70.213 (1.104) | 71.035 (1.116) | 69.505 (1.150) | 70.081 (1.099)
  Week 24 | 66.168 (1.184) | 70.884 (1.180) | 68.756 (1.193) | 70.454 (1.228) | 69.259 (1.174)

29. Secondary Outcome: 36-item-health Survey (SF-36) - General Mental Health Domain Score
Description: The 36-item-health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions evaluating patient's physical and mental health. Among the 36 questions, 1 is on the health comparing to 1 year ago and the remaining 35 questions are divided into 8 domains: Physical function, role limitations physical, Bodily pain, General physical health, Vitality, Social functioning, role limitations emotional, and General mental health.
  The domain score of general mental health (based on 5 questions) is reported, which is the weighted sum of the questions in the corresponding domain with the domain score ranging from 0 to 100. The higher the domain score, the better the mental health in general.
Time Frame: At Week 4, 12, and 24.
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 410 | 413 | 404 | 379 | 417
Score on a scale
  Week 4 | 69.585 (0.649) | 71.056 (0.646) | 70.927 (0.653) | 71.038 (0.674) | 71.281 (0.643)
  Week 12 | 69.201 (0.743) | 70.320 (0.740) | 70.362 (0.748) | 71.466 (0.772) | 71.048 (0.737)
  Week 24 | 68.144 (0.758) | 70.012 (0.755) | 69.868 (0.764) | 70.904 (0.788) | 69.286 (0.752)

30. Secondary Outcome: Number of Patients With at Least One Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Number of patients with at least one Chronic Obstructive Pulmonary Disease (COPD) exacerbation is reported. Incidence rate of Chronic Obstructive Pulmonary Disease (COPD) exacerbation is reported. A Chronic Obstructive Pulmonary Disease (COPD) exacerbation is defined as "a complex of lower respiratory events / symptoms (increase or new onset) related to the underlying COPD, with a duration of three days or more, requiring a change in treatment", where a "complex of lower respiratory events / symptoms" means at least two of the following: Shortness of breath, Sputum production (volume), Occurrence of purulent sputum, Cough, Wheezing, Chest tightness.
Time Frame: From first does until 30 days after the end of treatment, up to 205 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 429 | 419 | 415 | 390 | 427
Participants | 85 | 60 | 77 | 57 | 73

31. Secondary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Incidence rate of Chronic Obstructive Pulmonary Disease (COPD) exacerbation is reported. A Chronic Obstructive Pulmonary Disease (COPD) exacerbation is defined as "a complex of lower respiratory events / symptoms (increase or new onset) related to the underlying COPD, with a duration of three days or more, requiring a change in treatment", where a "complex of lower respiratory events / symptoms" means at least two of the following: Shortness of breath, Sputum production (volume), Occurrence of purulent sputum, Cough, Wheezing, Chest tightness.
Time Frame: From first does until 30 days after the end of treatment, up to 205 days.
Population: as for baseline characteristics
Measure: Number; unit: Events per patient-year
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
Number analyzed (Participants) | 429 | 419 | 415 | 390 | 427
Events per patient-year | 0.5797 | 0.4345 | 0.4898 | 0.4373 | 0.5332

ADVERSE EVENTS:
Time Frame: From first does until 30 days after the end of treatment, up to 205 days.
Description: Treated set: the treated set was defined as all patients who were randomized and who took at least one dose of trial medication.
Arm/Group | Placebo | BEA 2180 BR 50 Microgram (mcg) | BEA 2180 BR 100 Microgram (mcg) | BEA 2180 BR 200 Microgram (mcg) | Tiotropium Bromide 5 Microgram (mcg)
All-Cause Mortality (participants affected / at risk) | 5/429 | 3/419 | 3/415 | 7/390 | 2/427
Serious Adverse Events (participants affected / at risk) | 43/429 | 37/419 | 33/415 | 36/390 | 35/427
Other Adverse Events (participants affected / at risk) | 132/429 | 106/419 | 115/415 | 89/390 | 107/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=429) | BEA 2180 BR 50 Microgram (mcg) (N=419) | BEA 2180 BR 100 Microgram (mcg) (N=415) | BEA 2180 BR 200 Microgram (mcg) (N=390) | Tiotropium Bromide 5 Microgram (mcg) (N=427)
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dysthymic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 3 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 4 | 2
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Low cardiac output syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 2
Sudden death (General disorders) | 0 | 0 | 0 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 3 | 7 | 2 | 8
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 11 | 7 | 7 | 8
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tendon operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Aortic bypass (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=429) | BEA 2180 BR 50 Microgram (mcg) (N=419) | BEA 2180 BR 100 Microgram (mcg) (N=415) | BEA 2180 BR 200 Microgram (mcg) (N=390) | Tiotropium Bromide 5 Microgram (mcg) (N=427)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 85 | 60 | 66 | 53 | 68
Nasopharyngitis (Infections and infestations) | 38 | 28 | 33 | 27 | 27
Upper respiratory tract infection (Infections and infestations) | 20 | 26 | 21 | 13 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 15 | 14 | 11 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.